CLINICAL TRIAL: NCT03067623
Title: Intrauterine Infusion of Autologous Platelet-Rich Plasma (PRP) in Women With Thin Endometrium Undergoing Embryo-transfer.
Brief Title: Autologous Platelet-Rich Plasma (PRP) and Endometrial Thickness
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Roberta Venturella, Principal Investigator, University Magna Graecia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP-Et
Record Dates: First submitted 2017-02-26; First posted 2017-03-01 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Thin Endometrium; Endometrial Disorder; Endometrial Thickness Not Growing Under Estrogen Stimulation
Keywords: Thin endometrium; Endometrial thickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRP-infusion (Experimental): PRP will be obtained from a fresh whole blood collected from a peripheral vein; the blood sample will be centrifuged at 1500g (RCF) for 10 minutes and the repeated reversal of the tube will allow obtaining the PRP at the concentration required. Then 0,5-1ml of PRP will be infused into the uterine cavity through a Tomcat catheter. The endometrial thickening will be evaluated by ultrasonography 24-48h after the instillation and, if the endometrial lining reaches 7mm the Embryo-transfer will be arranged.
  Interventions: Drug: PRP; Device: Tomcat catheter

INTERVENTIONS:
Drug: PRP — PRP intrauterine infusion
Device: Tomcat catheter — PRP intrauterine infusion by means Tomcat catheter

SUMMARY:
The goal of this interventional study is to evaluate the increasing in endometrial thickening after the intrauterine infusion of 0,5-1 ml of autologous Platelet-Rich Plasma (PRP) and the implantation rate in women with thin endometrium undergoing Embryo-transfer, in order to propose a novel therapeutic approach for women with an endometrium < 7 mm unresponsive to standard treatments.

DETAILED DESCRIPTION:
In clinical practice, a thin endometrium, unresponsive to conventional therapies, usually results in cycle cancellation and embryo cryopreservation. The evaluation of an adequate endometrial growth is performed using grey-scale ultrasound. The minimal endometrial thickness required for embryo transfer is now considered about 7 mm at the end of natural or medically induced follicular phase, despite some investigators reported different cutoff values, ranging between 7 and 10 mm. Currently, no evidence-based data show the predictive positive value of endometrial thickness on pregnancy rate after Embryo-transfer, but if the endometrial lining is below 7mm the chance of pregnancy is statistically significant reduced.

Thin endometrium is relatively frequent in women with previous trauma of the uterus (cesarean sections, repetitive curettage), patients subjected to antitumoral treatments in childhood (Radiotherapy, Chemotherapy, Surgery), women affected by Asherman's syndrome, chronic infections (endometritis, Pelvic Inflammatory Disease) and inadequate blood flow (stress, malposition of uterus, fibrosis), patients with low estradiol values or excessive use of Clomiphene Citrate.

Several alternative treatments have been proposed over the years to improve the endometrial thickening, then showed themselves to be not considered the answer in many cases: some of them, indeed, require a not damaged endometrium, other act on endometrial blood flow and have no direct proliferative effect on the endometrium. The only factor presumed to have a proliferative effect on endometrium is the Granulocyte-Colony Stimulating Factor (G-CSF) but this hypothesis is not supported by in vitro studies.

Recently, first results from an in vitro study ongoing on the evaluation of Platelet-Rich Plasma (PRP) effect on endometrial cell proliferation have been presented (Aghayanova et al., 2016). The authors demonstrated that PRP increased proliferation not only on cultured fibroblasts, as currently known but also on mesenchymal cells, which are progenitors of different types of cells, including endometrial cells. This evidence supports the hypothesis that PRP stimulates some of the cellular processes involved in endometrial regeneration, that can be relevant to the management of a thin lining.

Autologous Platelet-Rich Plasma is prepared from fresh whole blood which is collected from a peripheral vein and processed to separate platelets from the other blood components. PRP contains activating platelets that stimulate the action of cytokines and growth factors. On the basis of this evidence, local intrauterine infusion of PRP may improve endometrial growth and implantation.

Patients considered to be candidates for a PRP application must undergo a minor hematological evaluation to exclude blood disorders or platelet dysfunction. The study, since it involves the use of a blood component, was approved by Ethical Committee and all participant have to sign an informed written consent before undergoing the procedure.

Any concerns of immunogenic reactions or disease transmission, that exist with homologous blood products, are eliminated because PRP is produced from autologous blood. Preparation of PRP, however, demands many processing steps, thus there is the theoretic possibility of contamination. For these reasons, all samples are subjected to quality and sterility controls within a closed mechanism. No wound infections after PRP applications have been reported. Despite PGF has mitogenic properties, there is no evidence that the growth factors included in PRP promote tumor growth or that they are involved in carcinogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial thickness < 7 mm under estrogen replacement therapy or repeated implantation failure
* Age between 18 and 46 years

Exclusion Criteria:

* Age < 18 and > 46 years
* Pregnancy
* Bleeding diathesis
* Previous uterine surgery (miomectomy, cesarean section, etc...)
* Platelet count < 105/μL
* Hemoglobin < 10 g/dL
* Presence of a tumor in the wound bed or metastatic disease
* Current diagnosis of cancer
* Other concomitant active infections

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 200 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-27 (Estimated)

PRIMARY OUTCOMES:
Endometrial thickness | 24-48h after the intrauterine PRP infusion
  Endometrial thickness > 7 mm measured by means of transvaginal ultrasound

SECONDARY OUTCOMES:
Positive pregnancy test rate | Approximately 3 weeks after treatment
  Positive pregnancy test rate after Embryo-transfer
Implantation rate | Approximately 6 weeks after treatment
  defined by number of gestational sacs seen on early pregnancy 6-week ultrasound divided by number of embryos transferred

OTHER OUTCOMES:
Clinical pregnancy rate | Approximately 8 weeks after treatment
  Defined by the number of fetal poles with heartbeat seen on 6-week ultrasound divided by the number of embryos transferred
Return to spontaneous period | Approximately 1 to 3 months after treatment
  Records of a menstrual flow diary (Menstrual Assessment Chart) for 1-3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Venturella, MD, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Pugliese Ciaccio Hospital, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang Y, Li J, Chen Y, Wei L, Yang X, Shi Y, Liang X. Autologous platelet-rich plasma promotes endometrial growth and improves pregnancy outcome during in vitro fertilization. Int J Clin Exp Med. 2015 Jan 15;8(1):1286-90. eCollection 2015. PMID 25785127
- [Background] Nazari L, Salehpour S, Hoseini S, Zadehmodarres S, Ajori L. Effects of autologous platelet-rich plasma on implantation and pregnancy in repeated implantation failure: A pilot study. Int J Reprod Biomed. 2016 Oct;14(10):625-628. PMID 27921085
- [Background] L. Aghajanova, S. Houshdaran, S. Balayan, J. Irwin, H. Huddleston, L. Giudice. Platelets for endometrial regeneration: a novel approach. Fertil Steril. Volume 106, Issue 3, Supplement, Page e82
- See also: Ongoing Trial — https://clinicaltrials.gov/ct2/show/record/NCT02825849?term=prp+endometrium&rank=2